CLINICAL TRIAL: NCT04030975
Title: Cognitive Process of Diagnostic Error in Emergency Physicians
Acronym: diagnosis
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Collaborators: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Cathay General Hosp. IRB, IRB, Cathay General Hospital
Other Study IDs: CGH-P103018; CGH-P103018 (Other: CGH)
Record Dates: First submitted 2014-05-27; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Thinking
Keywords: diagnostic error

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- interview: emergency physicians

SUMMARY:
Diagnostic error, Dual process model of reasoning) During the last decade, much emphasis has been placed on system solutions to patient safety problems. However, diagnostic error, despite being responsible for twice as many adverse events as medication error, has received little attention. The rate of diagnostic errors have been estimated to be between 0.6% to 12%.Some estimates are as high as 15%.The rate of negative outcome or adverse effects of diagnostic errors range from 6.9% to 17%. Most authors accept that the dual process model of reasoning explains how clinicians make diagnoses. The purpose of this study is to investigate why diagnostic errors occurred in the emergency departments (EDs).

DETAILED DESCRIPTION:
Diagnostic error, Dual process model of reasoning) During the last decade, much emphasis has been placed on system solutions to patient safety problems. However, diagnostic error, despite being responsible for twice as many adverse events as medication error, has received little attention. The rate of diagnostic errors have been estimated to be between 0.6% to 12%.Some estimates are as high as 15%.The rate of negative outcome or adverse effects of diagnostic errors range from 6.9% to 17%. Most authors accept that the dual process model of reasoning explains how clinicians make diagnoses. The purpose of this study is to investigate why diagnostic errors occurred in the emergency departments (EDs). A qualitative study approach was used with in-depth semi-structured interviews conducted with emergency physicians to investigate the cognitive diagnosis process. The study takes place in the EDs of three hospitals in Taiwan. We chose the participants using a purposive sampling technique to yield a sample that would be most likely contribute significant information on the diagnostic process. Sampling continued until novel information was no longer being gathered. All audiotapes were transcribed verbatim. The transcripts are analyzed by two of the investigators based on the ground theory. Once all relevant codes were identified, they were grouped together into meaningful categories. These categories were then grouped under appropriate themes, which were used to generate a theory of diagnostic errors.

ELIGIBILITY:
Inclusion Criteria:

* trained emergency physicians

Exclusion Criteria:

* refused interview

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: emergency physicians
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
generate a theory of diagnostic errors | Dec., 2015

CONTACTS AND LOCATIONS:
Overall Officials: Chaou-Shune Lin, MD, Principal Investigator — Hsinchu Cathay General Hospital
Locations (1):
- Cathay hospital, Taipei, Taiwan